CLINICAL TRIAL: NCT00349726
Title: Single-Dose Intravenous Inositol Pharmacokinetics in Preterm Infants
Acronym: INS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Eye Institute (NEI) (NIH); National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0036-1; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR025744 (NIH); UL1RR024979 (NIH)
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Retinopathy of Prematurity; Bronchopulmonary Dysplasia (BPD)
Keywords: NICHD Neonatal Research Network; Pharmacokinetics; Inositol; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity
MeSH Terms: conditions — Premature Birth; Retinopathy of Prematurity; Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Inositol low volume (Experimental): Single dose of intravenous inositol 5%, 60 mg/kg (1.2ml/kg) given over 20 minutes
  Interventions: Drug: Inositol lower volume
- Inositol high volume (Experimental): Single dose of intravenous inositol 5%, 120 mg/kg (2.4ml/kg) given over 20 minutes
  Interventions: Drug: Inositol higher volume
- Placebo low volume (Placebo Comparator): Placebo (5% glucose) at a volume equal to 60 mg/kg (1.2 ml/kg) given via IV over 20 minutes.
  Interventions: Drug: Placebo lower volume
- Placebo high volume (Placebo Comparator): Placebo (5% glucose) at a volume equal to 120 mg/kg (2.4 ml/kg) given via IV over 20 minutes
  Interventions: Drug: Placebo higher volume

INTERVENTIONS:
Drug: Inositol lower volume — 60 mg/kg (1.2ml/kg) of myo-inositol 5% given intravenously over 20 minutes.
  Arms: Inositol low volume
Drug: Inositol higher volume — 120 mg/kg (2.4ml/kg) of myo-inositol 5% given intravenously over 20 minutes.
  Arms: Inositol high volume
Drug: Placebo lower volume — 60 mg/kg (1.2ml/kg) of glucose 5% given intravenously over 20 minutes.
  Arms: Placebo low volume
Drug: Placebo higher volume — 120 mg/kg (2.4ml/kg) of glucose 5% given intravenously over 20 minutes.
  Arms: Placebo high volume

SUMMARY:
This pilot study was a randomized, placebo-controlled, clinical trial to measure changes in blood and urine levels of inositol in premature infants at high risk for retinopathy of prematurity (ROP) following a single intravenous dose of inositol. Based on previous studies, the premise is that maintaining inositol concentrations similar to those occurring naturally in utero will reduce the rates of ROP and bronchopulmonary dysplasia in premature infants. The objective was to evaluate the single-dose pharmacokinetics and safety of different amounts of intravenous myo-inositol (provided by Ross Products Division, Abbott Laboratories) in very low birth weight neonates, in preparation for a future Phase III multi-center randomized controlled trial. This study enrolled 74 infants at high risk for retinopathy at 9 NICHD Neonatal Research Network sites, and randomly assigned them to receive either 60mg/kg of 5% inositol, 120 mg/kg of 5% inositol, 60 mg/kg of 5% glucose (the placebo), or 120 mg/kg of 5% glucose.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is an abnormal growth of the blood vessels in the eye that occurs primarily in very premature infants. Eye development occurs normally in the womb; in infants born prematurely, however, the blood vessels must finish developing outside the protective environment of the uterus. Retinopathy of prematurity (also known as retrolental fibroplasia) is a leading cause of blindness and other vision impairments (myopia, strabismus, and amblyopia) in children, both in developed and developing countries.

Inositol is a naturally-occurring sugar alcohol produced by the placenta and is present in high levels in fetal blood throughout pregnancy in humans and other animals. Serum levels fall rapidly after birth, although this fall is moderated in infants who receive breast milk. Two randomized trials have shown that intravenous inositol supplementation in the first week significantly reduced death, bronchopulmonary dysplasia (BPD), and retinopathy. One study of oral supplements was less convincing, but also supported reduction of retinopathy.

This pilot study evaluated the half-life pharmacokinetics of a single-dose of myo-inositol (provided by Ross Products Division, Abbott Laboratories) in very low birth weight infants, looking at changes in blood and urine inositol levels. The premise is that maintaining inositol concentrations similar to those occurring naturally in utero will reduce the rates of retinopathy and bronchopulmonary dysplasia in premature infants. Results from this study will be used to select the doses for a subsequent multi-dose pilot study, and for the planned large multi-center trials.

In this study, nine NICHD Neonatal Research Network sites enrolled 74 infants of less than 30 weeks gestation and randomly assigned them to receive either 60mg/kg of 5% inositol, 120 mg/kg of 5% inositol, 60 mg/kg of 5% glucose (the placebo), or 120 mg/kg of 5% glucose. Concentrations of inositol were measured in both blood and urine to determine population pharmacokinetic parameters for these infants.

Stratification: Enrolled infants were stratified by age with 37 infants of 23 0/7 to 26 6/7 weeks in one group and 37 infants of 27 0/7 to 29 6/7 weeks in a second group.

ELIGIBILITY:
Inclusion Criteria:

* 23 0/7 to 26 6/7 weeks gestational age (36 infants) or
* 27 0/7 to 29 6/7 weeks gestational age (36 infants)
* 600-1500 grams birth weight
* No enteral feedings since birth at enrollment
* 3-6 days (25-132 hours) postnatal age

Note: Because of the high mortality expected in this population (15-20%), the study design (originally for 72 infants) required recruitment of a replacement subject if any infant failed to complete the four blood samples during the first week of the study.

Exclusion Criteria:

* Major congenital anomalies
* Moribund or not to be provided continued support
* Renal failure suspected (creatinine >2.5 with oliguria)
* Exchange transfusion received or expected to receive

Ages: 3 Days to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Population pharmacokinetics | 0-100 hours following infusion

SECONDARY OUTCOMES:
Adverse events during and following infusion, using a neonatal toxicity classification | Until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Roger G. Faix, MD, Principal Investigator — University of Utah; Barbara J. Stoll, MD, Principal Investigator — Emory University; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Ivan D. Frantz, III, MD, Principal Investigator — Tufts Medical Center
Locations (11):
- United States (11):
  - Yale University, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/